CLINICAL TRIAL: NCT05340699
Title: Safety and Efficacy of Defocus Distributed Multi-point Lens in Myopia Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY202003
Record Dates: First submitted 2022-03-22; First posted 2022-04-22 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): A group of children wearing Xingyouxue Defocus Distributed Multi-point lens
  Interventions: Device: Defocus Distributed Multi-point lens
- control group (Active Comparator): A group of children wearing single vision lens
  Interventions: Device: Single vision lens

INTERVENTIONS:
Device: Defocus Distributed Multi-point lens — Wear DDM lens
  Arms: experimental group
Device: Single vision lens — Wear single vision lens
  Arms: control group

SUMMARY:
Evaluate the safety and effectiveness of experimental group by comparing with the control group

DETAILED DESCRIPTION:
Compared the experimental group with the control group,the safety and effectiveness of DDM lens in mtopia control will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-13,with written consent of his/her guardian,regardless of gender;
* Objective cycloplegic spherical equivalent refractive between -1.00D and 5.00D,and best corrected vision acuity of right and left eyes are better than or equal to 1.0;
* Astigmatism less than or equal to -1.50D;
* Voluntarily participate in the clinical trial and sign the informed consent.

Exclusion Criteria:

* Those with a history of ocular trauma or intraocular surgery;
* Clinical significant slit-lamp findings;
* Abnormal IOP(<10 mmHg , >21 mmHg or difference between two eyes >5mmHg);
* Patient with other eye diseases,such as uveitis and other inflammation,glaucoma,cataract,fundus disease,eye tumors,eye trauma,strabismus and any lesions that affect vision function;
* Patient with systemic diseases causing immunosuppression,such as acute or chronic sinusitis,diabetes,Down syndrome,rheumatoid arthritis,psychosis and other conditions that the investigator considers inappropriate for wearing glasses;
* Those who have participated in other drug clinical trials within 3 months;
* Only one eye meets the inclusion criteria;
* Those who cannot have regular eye examinations;
* Those who have been involved in any myopia control clinical trials,previously used or are using RGP,contact lens and glasses or atropine drugs to control myopia in the past year;
* The candidates determined by the investigator are not eligible.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Objective cycloplegic refractive | baseline, 12 months
  Changes in objective cycloplegic refractive from baseline between two groups
Changes in Axial Length | baseline, 12 months
  Changes in axial length from baseline between two groups

SECONDARY OUTCOMES:
Changes in Objective cycloplegic refractive | baseline, 6 months，18 months and 24 months
  Changes in objective cycloplegic refractive from baseline between two groups
Changes in Axial length | baseline, 6 months，18 months and 24 months
  Changes in axial length from baseline between two groups
Changes in amplitude of accommodation | baseline, 6 months，18 months and 24 months
  Changes in amplitude of accommodation between two groups evey 6 months
Changes in near point of convergence | baseline, 6 months，18 months and 24 months
  Changes in near point of convergence between two groups evey 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqin Chen, MD, Principal Investigator — Tianjin Eye Hospital, Tianjin,China
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

REFERENCES:
- [Derived] Chen X, Li M, Li J, Wu M, Liu X, Yu C, Guo X, Wang Y, Wang Y, Lu W, Li L, Wang Y. One-year efficacy of myopia control by the defocus distributed multipoint lens: a multicentric randomised controlled trial. Br J Ophthalmol. 2024 Oct 22;108(11):1583-1589. doi: 10.1136/bjo-2023-324243. PMID 38503477